CLINICAL TRIAL: NCT00071383
Title: Analysis of Brain Metastasis in Patients With Breast Cancer, With and Without Over-Expression of HER-2
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040005; 04-N-0005
Record Dates: First submitted 2003-10-20; First posted 2003-10-13 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-11

CONDITIONS: Breast Neoplasms
Keywords: Herceptin; Trastuzumab; Microdissection; Proteomics; Microarrays; Metastatic Brain Tumor; Breast Cancer; Brain; Carcinoma; Genomics; Metastatic Breast Cancer; Metastatic Breast Tumor
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Carcinoma

SUMMARY:
This study will examine two subsets of patients with breast cancer metastasis, that is, spreading, to the brain. It will identify genes and proteins that promote metastasis, particularly in women who are found to over-express (have more than other people do) the human epidermal growth factor receptor, ErbB2, also known as HER-2. The molecular and genetic events that permit tumor metastasis are not well understood. There is intense investigation going on into the process in which tumor cells escape the primary local tumor, spread to distant places in the body, and find and create conditions that promote growth in those tissues. Metastasis of tumors such as breast cancer to the brain is a common problem. Tumor cells will be analyzed with the use of microarrays. A microarray is a tool for analyzing gene expression, consisting of a small membrane or glass slide containing samples of many genes arranged in a regular pattern. The goal is to identify a potential molecular signature. It is hoped that there will be discovery of why some patients are more likely than others to develop a brain metastasis, which can have a major negative effect on the quality of life and survival.

Female patients 18 years of age with known or evidence by radiology of a breast tumor metastatic to the brain or those who have had a removal of a brain tumor for diagnosis or treatment may be eligible for this study.

Participants will undergo the following procedures and tests:

* Craniotomy, that is, surgical opening of the skull, and removal of the brain tumor.
* Blood specimens taken from a central vein or artery before the operation, throughout as needed, and for several days afterward, to measure blood chemistries, blood count, and so forth.
* Physical examination and imaging of the central nervous system before and after surgery.
* Urine or serum, or both, pregnancy test of women of childbearing potential.

Patients will also undergo blood tests at 3-month intervals after surgery for up to 5 years. The purpose is to determine if there are tumor cells in the blood, which may explain how they reached the brain.

DETAILED DESCRIPTION:
Introduction: The molecular and genetic events that permit tumor metastasis are not well understood. The process whereby tumor cells escape the primary, local tumor, spread to distant sites in the body and find and create conditions conducive to growth in these disparate tissues remains an area of intense investigation. Metastasis of epithelial tumors, such as breast cancer, to the brain is a common problem, with significant consequences with respect to neurological dysfunction and shortening of survival.

Objective: To study two subset of patients with breast cancer metastatic to the brain, to identify genes and proteins that facilitate metastasis, particularly in women who over-express the growth factor receptor HER2, in which an increased risk of brain metastasis has recently been identified.

Study Population: 78 patients with breast cancer metastatic to the brain (39 women whose tumors are HER2-(-) and 39 women whose tumors are HER2-(+)) to compare with published microarray studies of non-metastatic breast cancer patients with these tumor types as well as with one another to help explain the differential trend toward metastasis in patients treated with Herceptin, a new therapy directed at HER-2 over-expressing tumors.

Anticipated Risks and Benefits: Less than minimal risk to the patients to sample tissue already removed from the brain as part of medically-necessary surgery and to sample blood. No direct benefit to the patient is expected.

Outcome Estimate and Potential Meaning for the Field: That this very detailed investigation of the genes and proteins expressed differentially between the non-metastatic and metastatic breast cancers, as well as between HER2-(-) and HER2-(+) subtypes will identify new or previously-unsuspected targets for new therapies to either prevent the development of brain metastasis or to treat these brain metastases more effectively.

ELIGIBILITY:
Inclusion Criteria:

1. A woman with a known or with radiographic evidence of a breast neoplasm metastatic to the brain.
2. Medically-indicated (diagnostic and/or therapeutic) brain tumor resection.
3. Informed consent from female patient, age 18 or older. In general, patients less than 18 years of age rarely have breast cancer metastatic to the brain.

Exclusion Criteria:

1. Inability to provide informed consent prior to surgery.
2. Medical conditions that cannot be corrected prior to surgery that would be standard contraindications for craniotomy (brain tumor patients).
3. Men.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78
Dates: Start 2003-10; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sorlie T, Tibshirani R, Parker J, Hastie T, Marron JS, Nobel A, Deng S, Johnsen H, Pesich R, Geisler S, Demeter J, Perou CM, Lonning PE, Brown PO, Borresen-Dale AL, Botstein D. Repeated observation of breast tumor subtypes in independent gene expression data sets. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8418-23. doi: 10.1073/pnas.0932692100. Epub 2003 Jun 26. PMID 12829800
- [Background] Pollack JR, Sorlie T, Perou CM, Rees CA, Jeffrey SS, Lonning PE, Tibshirani R, Botstein D, Borresen-Dale AL, Brown PO. Microarray analysis reveals a major direct role of DNA copy number alteration in the transcriptional program of human breast tumors. Proc Natl Acad Sci U S A. 2002 Oct 1;99(20):12963-8. doi: 10.1073/pnas.162471999. Epub 2002 Sep 24. PMID 12297621
- [Background] Sorlie T, Perou CM, Tibshirani R, Aas T, Geisler S, Johnsen H, Hastie T, Eisen MB, van de Rijn M, Jeffrey SS, Thorsen T, Quist H, Matese JC, Brown PO, Botstein D, Lonning PE, Borresen-Dale AL. Gene expression patterns of breast carcinomas distinguish tumor subclasses with clinical implications. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10869-74. doi: 10.1073/pnas.191367098. PMID 11553815